CLINICAL TRIAL: NCT02302066
Title: A Phase II, Double-Blind, Controlled Trial to Assess the Safety and Immunogenicity of Different Schedules of Takeda's Tetravalent Dengue Vaccine Candidate (TDV) in Healthy Subjects Aged Between 2 and <18 Years and Living in Dengue Endemic Countries in Asia and Latin America
Brief Title: Safety and Immunogenicity of Different Schedules of Takeda's Tetravalent Dengue Vaccine Candidate (TDV) in Healthy Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DEN-204; PHRR140804-000219 (Registry Identifier: PHRR); U1111-1154-2475 (Registry Identifier: WHO); 2018-003978-28 (Registry Identifier: EudraCT)
Record Dates: First submitted 2014-11-24; First posted 2014-11-26 (Estimated); Results first posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Dengue Fever
Keywords: Drug therapy
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (TDV 2-Dose) (Experimental): Takeda's tetravalent dengue vaccine candidate (TDV), 0.5 mL, subcutaneous injection on Days 1 and 91. Placebo-matching vaccine, 0.5 mL, subcutaneous injection on Day 365.
  Interventions: Biological: Takeda's Tetravalent Dengue Vaccine Candidate (TDV); Biological: TDV Placebo
- Group 2 (TDV 1-Dose) (Experimental): Takeda's tetravalent dengue vaccine candidate (TDV), 0.5 mL, subcutaneous injection on Day 1. Placebo-matching vaccine, 0.5 mL, subcutaneous injection on Days 91 and 365.
  Interventions: Biological: Takeda's Tetravalent Dengue Vaccine Candidate (TDV); Biological: TDV Placebo
- Group 3 (TDV 1-Dose + Booster) (Experimental): Takeda's tetravalent dengue vaccine candidate (TDV), 0.5 mL, subcutaneous injection on Days 1 and 365. Placebo-matching vaccine, 0.5 mL, subcutaneous injection on Day 91.
  Interventions: Biological: Takeda's Tetravalent Dengue Vaccine Candidate (TDV); Biological: TDV Placebo
- Group 4 (Placebo Control) (Placebo Comparator): Placebo-matching vaccine, 0.5 mL, subcutaneous injection on Days 1, 91 and 365.
  Interventions: Biological: TDV Placebo

INTERVENTIONS:
Biological: Takeda's Tetravalent Dengue Vaccine Candidate (TDV) — TDV subcutaneous injection
  Arms: Group 1 (TDV 2-Dose); Group 2 (TDV 1-Dose); Group 3 (TDV 1-Dose + Booster)
Biological: TDV Placebo — Placebo-matching vaccine

SUMMARY:
The purpose of this study is to assess the humoral immune responses to three different dose schedules of Takeda's Tetravalent Dengue Vaccine Candidate (TDV) administered subcutaneously in healthy participants between 2 and <18 years of age living in dengue endemic countries.

DETAILED DESCRIPTION:
The vaccine tested in this study is Takeda's Tetravalent Dengue Vaccine Candidate (TDV) which was administered in 3 different dosing schedules to participants aged from 2 to 17 years resident in dengue endemic countries. This study looked at the titers of antibodies to dengue fever elicited in people who received TDV.

The study randomized 1800 healthy participants. Participants were randomly assigned to one of the four treatment groups in a 1:2:5:1 ratio-which remained undisclosed to the participant and study doctor during the study (unless there was an urgent medical need):

* Group 1 - TDV 0.5 mL subcutaneous (SC) injection Days 1 and 91
* Group 2 - TDV 0.5 mL SC injection Day 1
* Group 3 - TDV 0.5 mL SC injection Days 1 and 365
* Group 4 - Placebo (dummy SC) - this is a liquid that looks like the study drug but has no active ingredient

A total of 600 participants were planned to be randomly included in immunogenicity analyses (approximately 100 participants planned in each of Group 1 and Group 4, and 200 participants planned in each of Group 2 and Group 3).

In order to keep the treatment arms undisclosed to the participant and the doctor, participants received a placebo injection at any study visit where TDV was not being administered (Days 1 and/or 91 and/or 365).

Participants were asked to record any symptoms that may be related to the vaccine or the injection site in a diary card for 28 days after each vaccination.

This multi-center trial was conducted in Asia and Latin America. Participants were followed for 48 months with 10 protocol-scheduled visits for participants included in the planned immunogenicity subset of approximately 600 subjects and 7 protocol-scheduled visits for subjects not included in the immunogenicity subset.

ELIGIBILITY:
Inclusion Criteria:

1. Is aged 2 to <18 years, at the time of enrolment.
2. Is in good health at the time of entry into the trial as determined by medical history, physical examination (including vital signs), and clinical judgment of the investigator.
3. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form (and assent form, where required) and any required privacy authorization prior to the initiation of any trial procedures, after the nature of the trial has been explained according to local regulatory requirements.
4. Can comply with trial procedures and are available for the duration of follow-up.

Exclusion Criteria:

1. Febrile illness (temperature ≥ 38°C or 100.4°F) or moderate or severe acute illness or infection at the time of enrolment. Trial entry should be delayed until the illness has improved.
2. Individuals with history or any illness that, in the opinion of the investigator, might interfere with the results of the trial or pose additional risk to the participants due to participation in the trial, including but not limited to: a. Known hypersensitivity or allergy to any of the vaccine components; b. Female participants who are pregnant or breastfeeding; c. Individuals with any serious chronic or progressive disease according to judgment of the investigator (e.g. neoplasm, insulin-dependent diabetes, cardiac, renal or hepatic disease, neurologic or seizure disorder or Guillain-Barré syndrome); d. Known or suspected impairment/alteration of immune function, including: i. Chronic use of oral steroids (Equivalent to 20 mg/day prednisone ≥ 12 weeks / ≥ 2 mg/kg body weight / day prednisone ≥ 2 weeks) within 60 days prior to Day 1 (use of inhaled, intranasal, or topical corticosteroids is allowed); ii. Receipt of parenteral steroids (Equivalent to 20 mg/day prednisone ≥ 12 weeks / ≥ 2 mg/kg body weight / day prednisone ≥ 2 weeks) within 60 days prior to Day 1; iii. Administration of immunoglobulins and/or any blood products within the three months preceding the first administration of the investigational vaccine or planned administration during the trial; iv. Receipt of immunostimulants within 60 days prior to Day 1; v. Immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within 6 months preceding (first) vaccination; vi. Human immunodeficiency virus (HIV) infection or HIV-related disease; vii. Genetic immunodeficiency.
3. Individuals who received any other vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrollment in this trial or who are planning to receive any vaccine within 28 days of investigational vaccine administration.
4. Individuals participating in any clinical trial with another investigational product 30 days prior to first trial visit or intent to participate in another clinical trial at any time during the conduct of this trial.
5. Individuals who are first degree relatives of individuals involved in trial conduct.
6. If female of childbearing potential, sexually active, and has not used any of the "acceptable contraceptive methods" for at least 2 months prior to trial entry: a. Of childbearing potential is defined as status post onset of menarche and not meeting any of the following conditions: menopausal (for at least 2 years), bilateral tubal ligation (at least 1 year previously), bilateral oophorectomy (at least 1 year previously) or hysterectomy; b. Acceptable birth control methods are defined as one or more of the following: i. Hormonal contraceptive (such as oral, injection, transdermal patch, implant, cervical ring); ii. Barrier (condom with spermicide or diaphragm with spermicide) each and every time during intercourse; iii. Intrauterine device (IUD); iv. Monogamous relationship with vasectomized partner. Partner must have been vasectomized for at least six months prior to the participants' trial entry.
7. If female of childbearing potential, sexually active and refuses to use an "acceptable contraceptive method" through to 6 weeks after the last dose of investigational vaccine.
8. Individuals who participated in a previous dengue vaccine trial.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1800 (Actual)
Dates: Start 2014-12-05 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2019-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Program Medical Director, Study Director — Takeda
Locations (3):
- Hospital Maternidad Nuestra Senora de la Altagracia, Santo Domingo, Distrito Nacional Santo Domingo, Dominican Republic
- Centro De Vacunacion Internacional, S.A.(CEVAXIN), Panama City, Panama
- Dela Salle Health Sciences Institute, Dasmariñas, Cavite, Philippines

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient/subject-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Rauscher M, Youard Z, Faccin A, Patel SS, Pang H, Zent O. Pregnancy outcomes following unintentional exposure to TAK-003, a live-attenuated tetravalent dengue vaccine. Expert Rev Vaccines. 2025 Dec;24(1):221-229. doi: 10.1080/14760584.2025.2480297. Epub 2025 Mar 27. PMID 40099800
- [Derived] Tricou V, Gottardo R, Egan MA, Clement F, Leroux-Roels G, Saez-Llorens X, Borkowski A, Wallace D, Dean HJ. Characterization of the cell-mediated immune response to Takeda's live-attenuated tetravalent dengue vaccine in adolescents participating in a phase 2 randomized controlled trial conducted in a dengue-endemic setting. Vaccine. 2022 Feb 16;40(8):1143-1151. doi: 10.1016/j.vaccine.2022.01.016. Epub 2022 Jan 22. PMID 35078666
- [Derived] Tsuji I, Dominguez D, Egan MA, Dean HJ. Development of a Novel Assay to Assess the Avidity of Dengue Virus-Specific Antibodies Elicited in Response to a Tetravalent Dengue Vaccine. J Infect Dis. 2022 May 4;225(9):1533-1544. doi: 10.1093/infdis/jiab064. PMID 33534885
- [Derived] Tricou V, Saez-Llorens X, Yu D, Rivera L, Jimeno J, Villarreal AC, Dato E, Saldana de Suman O, Montenegro N, DeAntonio R, Mazara S, Vargas M, Mendoza D, Rauscher M, Brose M, Lefevre I, Tuboi S, Borkowski A, Wallace D. Safety and immunogenicity of a tetravalent dengue vaccine in children aged 2-17 years: a randomised, placebo-controlled, phase 2 trial. Lancet. 2020 May 2;395(10234):1434-1443. doi: 10.1016/S0140-6736(20)30556-0. Epub 2020 Mar 17. PMID 32197107
- [Derived] Saez-Llorens X, Tricou V, Yu D, Rivera L, Jimeno J, Villarreal AC, Dato E, Mazara S, Vargas M, Brose M, Rauscher M, Tuboi S, Borkowski A, Wallace D. Immunogenicity and safety of one versus two doses of tetravalent dengue vaccine in healthy children aged 2-17 years in Asia and Latin America: 18-month interim data from a phase 2, randomised, placebo-controlled study. Lancet Infect Dis. 2018 Feb;18(2):162-170. doi: 10.1016/S1473-3099(17)30632-1. Epub 2017 Nov 6. PMID 29122463
- [Derived] Saez-Llorens X, Tricou V, Yu D, Rivera L, Tuboi S, Garbes P, Borkowski A, Wallace D. Safety and immunogenicity of one versus two doses of Takeda's tetravalent dengue vaccine in children in Asia and Latin America: interim results from a phase 2, randomised, placebo-controlled study. Lancet Infect Dis. 2017 Jun;17(6):615-625. doi: 10.1016/S1473-3099(17)30166-4. Epub 2017 Mar 30. PMID 28365225

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 3 investigative sites in Dominican Republic, Panama and Philippines from 05 Dec 2014 to 18 Feb 2019.
Pre-assignment Details: Healthy volunteers were enrolled in a 1:2:5:1 ratio into 4 study groups: Group 1 received two doses of Tetravalent Dengue Vaccine (TDV), Group 2 received one dose of TDV, Group 3 received one dose of TDV along with booster vaccination and Group 4 received placebo.
Groups:
- Group 1 (TDV 2-Dose): Takeda's tetravalent dengue vaccine candidate (TDV), 0.5 mL, subcutaneous injection on Days 1 and 91. Placebo-matching, 0.5 mL, subcutaneous injection on Day 365.
- Group 2 (TDV 1-Dose): Takeda's TDV, 0.5 mL, subcutaneous injection on Day 1. Placebo-matching, 0.5 mL, subcutaneous injection on Days 91 and 365.
- Group 3 (TDV 1-Dose + Booster): Takeda's TDV, 0.5 mL, subcutaneous injection on Days 1 and 365. Placebo-matching, 0.5 mL, subcutaneous injection on Day 91.
- Group 4 (Placebo Control): Placebo-matching, 0.5 mL, subcutaneous injection on Days 1, 91 and 365.
Period: Overall Study
Arm/Group | Group 1 (TDV 2-Dose) | Group 2 (TDV 1-Dose) | Group 3 (TDV 1-Dose + Booster) | Group 4 (Placebo Control)
Started | 201 | 398 | 1002 | 199
Safety Analysis Set | 200 | 398 | 998 | 198
Immunogenicity Subset | 92 | 187 | 192 | 94
Per-Protocol Set (PPS) | 83 | 171 | 174 | 81
Completed | 168 | 323 | 830 | 158
Not Completed | 33 | 75 | 172 | 41
Not completed — Adverse Event | 1 | 1 | 3 | 0
Not completed — Lost to Follow-up | 4 | 5 | 24 | 7
Not completed — Withdrawal by Subject | 25 | 58 | 124 | 33
Not completed — Pregnancy | 2 | 10 | 12 | 0
Not completed — Reason Not Specified | 1 | 1 | 9 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who received at least 1 dose of trial vaccine.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (TDV 2-Dose) | Group 2 (TDV 1-Dose) | Group 3 (TDV 1-Dose + Booster) | Group 4 (Placebo Control) | Total
Number analyzed (Participants) | 200 | 398 | 998 | 198 | 1794
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.3 (4.01) | 7.3 (4.14) | 7.3 (4.06) | 7.0 (3.96) | 7.3 (4.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 207 | 486 | 95 | 888
  Male | 100 | 191 | 512 | 103 | 906
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 165 | 317 | 825 | 158 | 1465
  Not Hispanic or Latino | 35 | 81 | 173 | 40 | 329
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 102 | 204 | 505 | 101 | 912
  Asian | 35 | 82 | 174 | 40 | 331
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 63 | 110 | 311 | 56 | 540
  White | 0 | 2 | 8 | 1 | 11
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] | 122.1 (22.59) | 120.9 (23.15) | 121.4 (22.60) | 119.3 (21.88) | 121.2 (22.64)
Weight [Mean (Standard Deviation); unit: kg] | 27.86 (15.069) | 27.25 (14.368) | 27.12 (13.612) | 25.66 (13.371) | 27.07 (13.924)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index=weight/[height^2]
  kg/m^2 | 17.42 (3.558) | 17.43 (3.306) | 17.29 (3.123) | 16.93 (2.975) | 17.30 (3.200)

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Neutralizing Antibodies (Microneutralization Test [MNT50]) for Each of the Four DENV Serotypes for Participants in the Immunogenicity Subset
Description: GMTs of neutralizing antibodies were measured by microneutralization test 50% [MNT50] for each of the 4 Dengue Serotypes. The 4 dengue virus serotypes were DENV-1, DENV-2, DENV-3 and DENV-4. Data reported for up to Month 48 was collected at Months 1, 3, 6, 12, 13, 18, 24, 36 and 48.
Time Frame: Up to Month 48
Population: Per Protocol Set (PPS): All participants who received at least 1 dose of trial vaccine, who had a valid pre-dose and at least 1 valid post-dose measurement for immunogenicity and no major protocol violations. PPS included only participants from Immunogenicity Subset. Number analyzed are participants with data available at the given timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1 (TDV 2-Dose) | Group 2 (TDV 1-Dose) | Group 3 (TDV 1-Dose + Booster) | Group 4 (Placebo Control)
Number analyzed (Participants) | 83 | 171 | 174 | 81
titer
  DENV-1, Day 28 (Month 1) | 768.2 [498.7 to 1183.4] | 999.7 [723.6 to 1381.2] | 920.9 [689.4 to 1230.1] | 60.7 [31.8 to 116.0]
  DENV-2, Day 28 (Month 1) | 4329.7 [2847.6 to 6583.2] | 4219.3 [3118.9 to 5708.1] | 3572.2 [2674.6 to 4771.2] | 75.0 [39.6 to 141.8]
  DENV-3, Day 28 (Month 1) | 216.1 [124.7 to 374.6] | 352.8 [237.5 to 524.2] | 363.6 [249.8 to 529.1] | 45.8 [25.9 to 81.1]
  DENV-4, Day 28 (Month 1) | 199.2 [130.0 to 305.2] | 317.3 [232.2 to 433.5] | 260.4 [195.0 to 347.7] | 24.8 [16.2 to 38.0]
  DENV-1, Day 91 (Month 3) | 422.3 [256.7 to 695.0] | 684.2 [491.4 to 952.8] | 708.9 [522.6 to 961.6] | 64.6 [33.8 to 123.4]
  DENV-2, Day 91 (Month 3) | 1810.1 [1311.1 to 2499.2] | 2216.9 [1750.8 to 2807.2] | 1709.6 [1370.4 to 2132.7] | 76.0 [40.1 to 144.3]
  DENV-3, Day 91 (Month 3) | 140.8 [83.8 to 236.6] | 250.8 [174.5 to 360.6] | 251.9 [175.7 to 361.2] | 39.3 [22.6 to 68.2]
  DENV-4, Day 91 (Month 3) | 122.9 [77.6 to 194.6] | 170.8 [122.6 to 237.8] | 147.0 [108.4 to 199.2] | 23.4 [14.9 to 36.9]
  DENV-1, Day 180 (Month 6): number analyzed (Participants) | 83 | 170 | 174 | 81
  DENV-1, Day 180 (Month 6) | 448.8 [293.0 to 687.5] | 463.7 [329.5 to 652.6] | 538.9 [391.2 to 742.3] | 55.7 [29.2 to 106.6]
  DENV-2, Day 180 (Month 6): number analyzed (Participants) | 83 | 170 | 174 | 81
  DENV-2, Day 180 (Month 6) | 1461.5 [1071.7 to 1992.9] | 1682.9 [1333.5 to 2124.0] | 1335.1 [1067.7 to 1669.5] | 77.2 [39.8 to 149.6]
  DENV-3, Day 180 (Month 6): number analyzed (Participants) | 83 | 170 | 174 | 81
  DENV-3, Day 180 (Month 6) | 150.1 [96.9 to 232.6] | 166.3 [117.6 to 235.3] | 173.9 [125.8 to 240.5] | 37.4 [21.7 to 64.6]
  DENV-4, Day 180 (Month 6): number analyzed (Participants) | 83 | 170 | 174 | 81
  DENV-4, Day 180 (Month 6) | 109.1 [72.9 to 163.2] | 110.0 [81.0 to 149.2] | 92.3 [68.7 to 123.9] | 22.3 [14.1 to 35.1]
  DENV-1, Day 365 (Month 12): number analyzed (Participants) | 79 | 161 | 164 | 76
  DENV-1, Day 365 (Month 12) | 370.7 [232.3 to 591.8] | 409.6 [287.9 to 582.5] | 487.3 [346.2 to 686.0] | 72.7 [38.0 to 139.1]
  DENV-2, Day 365 (Month 12): number analyzed (Participants) | 79 | 161 | 164 | 76
  DENV-2, Day 365 (Month 12) | 1070.0 [746.7 to 1533.2] | 1529.8 [1179.0 to 1985.0] | 1041.0 [802.8 to 1349.9] | 133.9 [67.7 to 264.9]
  DENV-3, Day 365 (Month 12): number analyzed (Participants) | 79 | 161 | 164 | 76
  DENV-3, Day 365 (Month 12) | 166.8 [101.4 to 274.2] | 201.0 [139.0 to 290.4] | 199.2 [138.7 to 286.1] | 62.0 [34.6 to 111.0]
  DENV-4, Day 365 (Month 12): number analyzed (Participants) | 79 | 161 | 164 | 76
  DENV-4, Day 365 (Month 12) | 87.9 [57.7 to 133.8] | 85.6 [63.0 to 116.3] | 89.3 [64.5 to 123.6] | 29.3 [18.5 to 46.6]
  DENV-1, Day 393 (Month 13): number analyzed (Participants) | 80 | 163 | 167 | 75
  DENV-1, Day 393 (Month 13) | 454.4 [273.4 to 755.2] | 385.8 [271.6 to 548.2] | 1598.8 [1258.2 to 2031.6] | 80.6 [41.4 to 156.9]
  DENV-2, Day 393 (Month 13): number analyzed (Participants) | 80 | 163 | 167 | 75
  DENV-2, Day 393 (Month 13) | 1152.4 [796.3 to 1667.6] | 1384.1 [1066.3 to 1796.7] | 1866.1 [1551.4 to 2244.6] | 129.5 [64.9 to 258.6]
  DENV-3, Day 393 (Month 13): number analyzed (Participants) | 80 | 163 | 167 | 75
  DENV-3, Day 393 (Month 13) | 192.1 [115.3 to 320.3] | 225.1 [157.1 to 322.7] | 767.6 [615.4 to 957.4] | 68.5 [36.5 to 128.8]
  DENV-4, Day 393 (Month 13): number analyzed (Participants) | 80 | 163 | 167 | 75
  DENV-4, Day 393 (Month 13) | 90.5 [58.1 to 141.2] | 86.3 [64.2 to 116.1] | 278.0 [226.6 to 340.9] | 28.8 [18.0 to 46.0]
  DENV-1, Day 540 (Month 18): number analyzed (Participants) | 81 | 168 | 172 | 80
  DENV-1, Day 540 (Month 18) | 475.9 [286.3 to 791.0] | 461.3 [329.1 to 646.6] | 1056.3 [804.0 to 1387.9] | 92.2 [49.1 to 172.9]
  DENV-2, Day 540 (Month 18): number analyzed (Participants) | 81 | 168 | 172 | 80
  DENV-2, Day 540 (Month 18) | 1211.5 [841.6 to 1744.1] | 1241.8 [947.1 to 1628.1] | 1456.6 [1181.7 to 1795.5] | 176.7 [92.8 to 336.7]
  DENV-3, Day 540 (Month 18): number analyzed (Participants) | 81 | 168 | 172 | 80
  DENV-3, Day 540 (Month 18) | 285.5 [170.7 to 477.5] | 298.0 [205.0 to 433.3] | 548.0 [411.2 to 730.3] | 77.6 [44.0 to 136.9]
  DENV-4, Day 540 (Month 18): number analyzed (Participants) | 81 | 168 | 172 | 80
  DENV-4, Day 540 (Month 18) | 98.3 [64.5 to 149.9] | 102.0 [75.1 to 138.6] | 171.6 [132.9 to 221.6] | 33.1 [21.1 to 51.9]
  DENV-1, Day 730 (Month 24): number analyzed (Participants) | 71 | 145 | 148 | 70
  DENV-1, Day 730 (Month 24) | 471.1 [289.9 to 765.4] | 441.5 [302.4 to 644.3] | 920.9 [699.9 to 1211.8] | 114.5 [58.8 to 223.0]
  DENV-2, Day 730 (Month 24): number analyzed (Participants) | 71 | 145 | 148 | 70
  DENV-2, Day 730 (Month 24) | 1395.5 [962.1 to 2024.3] | 1748.2 [1328.8 to 2300.0] | 1685.8 [1346.1 to 2111.3] | 244.6 [118.2 to 506.3]
  DENV-3, Day 730 (Month 24): number analyzed (Participants) | 71 | 145 | 148 | 70
  DENV-3, Day 730 (Month 24) | 243.0 [144.2 to 409.3] | 276.0 [188.3 to 404.7] | 470.1 [347.7 to 635.7] | 90.8 [46.6 to 176.8]
  DENV-4, Day 730 (Month 24): number analyzed (Participants) | 71 | 145 | 148 | 70
  DENV-4, Day 730 (Month 24) | 180.0 [113.5 to 285.6] | 170.4 [121.3 to 239.4] | 285.9 [219.6 to 372.1] | 56.3 [32.1 to 98.9]
  DENV-1, Day 1095 (Month 36): number analyzed (Participants) | 66 | 137 | 139 | 66
  DENV-1, Day 1095 (Month 36) | 495.2 [278.9 to 879.3] | 364.7 [246.3 to 540.1] | 742.8 [553.6 to 996.8] | 90.7 [47.3 to 173.7]
  DENV-2, Day 1095 (Month 36): number analyzed (Participants) | 66 | 137 | 139 | 66
  DENV-2, Day 1095 (Month 36) | 1394.2 [946.4 to 2053.9] | 1408.4 [1057.3 to 1876.0] | 1476.2 [1153.3 to 1889.7] | 203.5 [100.0 to 414.0]
  DENV-3, Day 1095 (Month 36): number analyzed (Participants) | 66 | 137 | 139 | 66
  DENV-3, Day 1095 (Month 36) | 262.8 [158.2 to 436.5] | 214.9 [144.5 to 319.7] | 364.8 [266.4 to 499.4] | 66.4 [35.1 to 125.5]
  DENV-4, Day 1095 (Month 36): number analyzed (Participants) | 66 | 137 | 139 | 66
  DENV-4, Day 1095 (Month 36) | 201.8 [125.2 to 325.3] | 148.1 [104.8 to 209.3] | 236.1 [179.4 to 310.6] | 45.7 [27.0 to 77.2]
  DENV-1, Day 1460 (Month 48): number analyzed (Participants) | 65 | 133 | 136 | 63
  DENV-1, Day 1460 (Month 48) | 377.8 [226.1 to 631.5] | 421.0 [285.1 to 621.9] | 718.5 [537.7 to 959.9] | 100.0 [49.8 to 200.7]
  DENV-2, Day 1460 (Month 48): number analyzed (Participants) | 65 | 133 | 136 | 63
  DENV-2, Day 1460 (Month 48) | 1051.9 [732.2 to 1511.1] | 1319.0 [970.1 to 1793.5] | 1200.0 [927.1 to 1553.1] | 208.1 [99.2 to 436.5]
  DENV-3, Day 1460 (Month 48): number analyzed (Participants) | 65 | 133 | 136 | 63
  DENV-3, Day 1460 (Month 48) | 183.4 [112.9 to 298.0] | 200.5 [135.1 to 297.6] | 287.5 [210.7 to 392.4] | 71.3 [36.6 to 138.9]
  DENV-4, Day 1460 (Month 48): number analyzed (Participants) | 65 | 133 | 136 | 63
  DENV-4, Day 1460 (Month 48) | 152.0 [96.6 to 239.2] | 164.1 [114.1 to 236.0] | 218.6 [164.7 to 290.2] | 46.2 [26.1 to 81.8]

2. Secondary Outcome: Seropositivity Rates For Each of the 4 Dengue Serotypes for Participants in the Immunogenicity Subset
Description: Seropositivity rate, defined as the percentage of participants seropositive, was derived from the titers of dengue-neutralizing antibodies. Seropositivity defined as a reciprocal neutralizing titer ≥10 (for each serotype). The 4 dengue virus serotypes were DENV-1, DENV-2, DENV-3 and DENV-4.
Time Frame: Months 1, 3, 6, 12, 13, 18, 24, 36, and 48
Population: PPS included all participants who received at least 1 dose of trial vaccine, who had a valid pre-dose and at least 1 valid post-dose measurement for immunogenicity and no major protocol violations. PPS included only participants from Immunogenicity Subset. Number analyzed are participants with data available at the given timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 (TDV 2-Dose) | Group 2 (TDV 1-Dose) | Group 3 (TDV 1-Dose + Booster) | Group 4 (Placebo Control)
Number analyzed (Participants) | 83 | 171 | 174 | 81
percentage of participants
  DENV-1, Day 28 (Month 1) | 97.6 [91.6 to 99.7] | 97.7 [94.1 to 99.4] | 100.0 [97.9 to 100.0] | 49.4 [38.1 to 60.7]
  DENV-2, Day 28 (Month 1) | 96.4 [89.8 to 99.2] | 95.3 [91.0 to 98.0] | 96.6 [92.6 to 98.7] | 51.9 [40.5 to 63.1]
  DENV-3, Day 28 (Month 1) | 88.0 [79.0 to 94.1] | 90.1 [84.6 to 94.1] | 90.8 [85.5 to 94.7] | 50.6 [39.3 to 61.9]
  DENV-4, Day 28 (Month 1) | 94.0 [86.5 to 98.0] | 93.6 [88.8 to 96.7] | 95.4 [91.1 to 98.0] | 49.4 [38.1 to 60.7]
  DENV-1, Day 91 (Month 3) | 95.2 [88.1 to 98.7] | 97.7 [94.1 to 99.4] | 99.4 [96.8 to 100.0] | 51.9 [40.5 to 63.1]
  DENV-2, Day 91 (Month 3) | 98.8 [93.5 to 100.0] | 98.8 [95.8 to 99.9] | 99.4 [96.8 to 100.0] | 53.1 [41.7 to 64.3]
  DENV-3, Day 91 (Month 3) | 89.2 [80.4 to 94.9] | 95.3 [91.0 to 98.0] | 91.4 [86.2 to 95.1] | 48.1 [36.9 to 59.5]
  DENV-4, Day 91 (Month 3) | 88.0 [79.0 to 94.1] | 90.6 [85.3 to 94.6] | 90.8 [85.5 to 94.7] | 45.7 [34.6 to 57.1]
  DENV-1, Day 180 (Month 6): number analyzed (Participants) | 83 | 170 | 174 | 81
  DENV-1, Day 180 (Month 6) | 100.0 [95.7 to 100.0] | 97.1 [93.3 to 99.0] | 99.4 [96.8 to 100.0] | 49.4 [38.1 to 60.7]
  DENV-2, Day 180 (Month 6): number analyzed (Participants) | 83 | 170 | 174 | 81
  DENV-2, Day 180 (Month 6) | 98.8 [93.5 to 100.0] | 99.4 [96.8 to 100.0] | 99.4 [96.8 to 100.0] | 49.4 [38.1 to 60.7]
  DENV-3, Day 180 (Month 6): number analyzed (Participants) | 83 | 170 | 174 | 81
  DENV-3, Day 180 (Month 6) | 98.8 [93.5 to 100.0] | 92.9 [88.0 to 96.3] | 93.1 [88.3 to 96.4] | 48.1 [36.9 to 59.5]
  DENV-4, Day 180 (Month 6): number analyzed (Participants) | 83 | 170 | 174 | 81
  DENV-4, Day 180 (Month 6) | 92.8 [84.9 to 97.3] | 90.6 [85.2 to 94.5] | 85.1 [78.9 to 90.0] | 44.4 [33.4 to 55.9]
  DENV-1, Day 365 (Month 12): number analyzed (Participants) | 79 | 161 | 164 | 76
  DENV-1, Day 365 (Month 12) | 98.7 [93.1 to 100.0] | 97.5 [93.8 to 99.3] | 97.6 [93.9 to 99.3] | 57.9 [46.0 to 69.1]
  DENV-2, Day 365 (Month 12): number analyzed (Participants) | 79 | 161 | 164 | 76
  DENV-2, Day 365 (Month 12) | 98.7 [93.1 to 100.0] | 99.4 [96.6 to 100.0] | 100.0 [97.8 to 100.0] | 60.5 [48.6 to 71.6]
  DENV-3, Day 365 (Month 12): number analyzed (Participants) | 79 | 161 | 164 | 76
  DENV-3, Day 365 (Month 12) | 94.9 [87.5 to 98.6] | 94.4 [89.7 to 97.4] | 90.2 [84.6 to 94.3] | 57.9 [46.0 to 69.1]
  DENV-4, Day 365 (Month 12): number analyzed (Participants) | 79 | 161 | 164 | 76
  DENV-4, Day 365 (Month 12) | 92.4 [84.2 to 97.2] | 85.1 [78.6 to 90.2] | 82.9 [76.3 to 88.3] | 55.3 [43.4 to 66.7]
  DENV-1, Day 393 (Month 13): number analyzed (Participants) | 80 | 163 | 167 | 75
  DENV-1, Day 393 (Month 13) | 97.5 [91.3 to 99.7] | 95.7 [91.4 to 98.3] | 100.0 [97.8 to 100.0] | 60.0 [48.0 to 71.1]
  DENV-2, Day 393 (Month 13): number analyzed (Participants) | 80 | 163 | 167 | 75
  DENV-2, Day 393 (Month 13) | 98.8 [93.2 to 100.0] | 98.8 [95.6 to 99.9] | 100.0 [97.8 to 100.0] | 61.3 [49.4 to 72.4]
  DENV-3, Day 393 (Month 13): number analyzed (Participants) | 80 | 163 | 167 | 75
  DENV-3, Day 393 (Month 13) | 95.0 [87.7 to 98.6] | 95.1 [90.6 to 97.9] | 100.0 [97.8 to 100.0] | 57.3 [45.4 to 68.7]
  DENV-4, Day 393 (Month 13): number analyzed (Participants) | 80 | 163 | 167 | 75
  DENV-4, Day 393 (Month 13) | 90.0 [81.2 to 95.6] | 86.5 [80.3 to 91.3] | 100.0 [97.8 to 100.0] | 53.3 [41.4 to 64.9]
  DENV-1, Day 540 (Month 18): number analyzed (Participants) | 81 | 168 | 172 | 80
  DENV-1, Day 540 (Month 18) | 95.1 [87.8 to 98.6] | 97.0 [93.2 to 99.0] | 98.8 [95.9 to 99.9] | 62.5 [51.0 to 73.1]
  DENV-2, Day 540 (Month 18): number analyzed (Participants) | 81 | 168 | 172 | 80
  DENV-2, Day 540 (Month 18) | 98.8 [93.3 to 100.0] | 97.6 [94.0 to 99.3] | 100.0 [97.9 to 100.0] | 68.8 [57.4 to 78.7]
  DENV-3, Day 540 (Month 18): number analyzed (Participants) | 81 | 168 | 172 | 80
  DENV-3, Day 540 (Month 18) | 95.1 [87.8 to 98.6] | 92.3 [87.1 to 95.8] | 98.3 [95.0 to 99.6] | 63.8 [52.2 to 74.2]
  DENV-4, Day 540 (Month 18): number analyzed (Participants) | 81 | 168 | 172 | 80
  DENV-4, Day 540 (Month 18) | 87.7 [78.5 to 93.9] | 86.9 [80.8 to 91.6] | 97.1 [93.3 to 99.0] | 57.5 [45.9 to 68.5]
  DENV-1, Day 730 (Month 24): number analyzed (Participants) | 71 | 145 | 148 | 70
  DENV-1, Day 730 (Month 24) | 100.0 [94.9 to 100.0] | 95.9 [91.2 to 98.5] | 100.0 [97.5 to 100.0] | 68.6 [56.4 to 79.1]
  DENV-2, Day 730 (Month 24): number analyzed (Participants) | 71 | 145 | 148 | 70
  DENV-2, Day 730 (Month 24) | 100.0 [94.9 to 100.0] | 99.3 [96.2 to 100.0] | 100.0 [97.5 to 100.0] | 71.4 [59.4 to 81.6]
  DENV-3, Day 730 (Month 24): number analyzed (Participants) | 71 | 145 | 148 | 70
  DENV-3, Day 730 (Month 24) | 94.4 [86.2 to 98.4] | 93.1 [87.7 to 96.6] | 98.6 [95.2 to 99.8] | 65.7 [53.4 to 76.7]
  DENV-4, Day 730 (Month 24): number analyzed (Participants) | 71 | 145 | 148 | 70
  DENV-4, Day 730 (Month 24) | 94.4 [86.2 to 98.4] | 91.7 [86.0 to 95.7] | 98.6 [95.2 to 99.8] | 61.4 [49.0 to 72.8]
  DENV-1, Day 1095 (Month 36): number analyzed (Participants) | 66 | 137 | 139 | 66
  DENV-1, Day 1095 (Month 36) | 100.0 [94.6 to 100.0] | 92.7 [87.0 to 96.4] | 100.0 [97.4 to 100.0] | 68.2 [55.6 to 79.1]
  DENV-2, Day 1095 (Month 36): number analyzed (Participants) | 66 | 137 | 139 | 66
  DENV-2, Day 1095 (Month 36) | 100.0 [94.6 to 100.0] | 99.3 [96.0 to 100.0] | 100.0 [97.4 to 100.0] | 71.2 [58.7 to 81.7]
  DENV-3, Day 1095 (Month 36): number analyzed (Participants) | 66 | 137 | 139 | 66
  DENV-3, Day 1095 (Month 36) | 97.0 [89.5 to 99.6] | 88.3 [81.7 to 93.2] | 98.6 [94.9 to 99.8] | 63.6 [50.9 to 75.1]
  DENV-4, Day 1095 (Month 36): number analyzed (Participants) | 66 | 137 | 139 | 66
  DENV-4, Day 1095 (Month 36) | 95.5 [87.3 to 99.1] | 88.3 [81.7 to 93.2] | 98.6 [94.9 to 99.8] | 63.6 [50.9 to 75.1]
  DENV-1, Day 1460 (Month 48): number analyzed (Participants) | 65 | 133 | 136 | 63
  DENV-1, Day 1460 (Month 48) | 96.9 [89.3 to 99.6] | 94.7 [89.5 to 97.9] | 100.0 [97.3 to 100.0] | 68.3 [55.3 to 79.4]
  DENV-2, Day 1460 (Month 48): number analyzed (Participants) | 65 | 133 | 136 | 63
  DENV-2, Day 1460 (Month 48) | 100.0 [94.5 to 100.0] | 98.5 [94.7 to 99.8] | 100.0 [97.3 to 100.0] | 68.3 [55.3 to 79.4]
  DENV-3, Day 1460 (Month 48): number analyzed (Participants) | 65 | 133 | 136 | 63
  DENV-3, Day 1460 (Month 48) | 95.4 [87.1 to 99.0] | 90.2 [83.9 to 94.7] | 97.8 [93.7 to 99.5] | 63.5 [50.4 to 75.3]
  DENV-4, Day 1460 (Month 48): number analyzed (Participants) | 65 | 133 | 136 | 63
  DENV-4, Day 1460 (Month 48) | 90.8 [81.0 to 96.5] | 91.0 [84.8 to 95.3] | 99.3 [96.0 to 100.0] | 60.3 [47.2 to 72.4]

3. Secondary Outcome: Percentage of Participants With Solicited Local (Injection Site) Adverse Events (AEs) (Diary Recorded) by Severity in the Immunogenicity Subset of Infant/Toddler Following Each Vaccination
Description: Solicited local injection included pain, erythema at injection site, and swelling at injection site. They were collected using a diary and graded as [Grade 0 (no pain), 1 (mild: minor reaction to touch), 2 (moderate: cries/protests on touch) and 3 (severe: cries when limb is moved/spontaneously painful)]. Erythema and Swelling at injection site were graded as Grade 0 (<10 mm), 1 (mild: ≥10 - ≤ 20 mm), 2 (moderate: > 20 - ≤ 40 mm) and 3 (severe: > 40 mm).
Time Frame: Within 7 days after each vaccination
Population: Safety Analysis Set included all participants who received at least 1 dose of trial vaccine. Only participants in immunogenicity subset were included. Data were summarized separately for each age group. Number analyzed are participants with data available for the category. Only categories for which there was at least 1 participant are reported.
Measure: Number; unit: percentage of participants
Groups:
- Group 1 (TDV 2-Dose) Infant/Toddler: Participants aged <6 years received Takeda's tetravalent dengue vaccine candidate (TDV), 0.5 mL, subcutaneous injection on Days 1 and 91. Placebo-matching, 0.5 mL, subcutaneous injection on Day 365.
- Group 2 (TDV 1-Dose) Infant/Toddler: Participants aged <6 years received Takeda's TDV, 0.5 mL, subcutaneous injection on Day 1. Placebo-matching, 0.5 mL, subcutaneous injection on Days 91 and 365.
- Group 3 (TDV 2-Dose) Infant/Toddler: Participants aged <6 years received Takeda's TDV, 0.5 mL, subcutaneous injection on Days 1 and 365. Placebo-matching, 0.5 mL, subcutaneous injection on Day 91.
- Group 4 (Placebo Control) Infant/Toddler: Participants aged <6 years received placebo-matching, 0.5 mL, subcutaneous injection on Days 1, 91 and 365.
Arm/Group | Group 1 (TDV 2-Dose) Infant/Toddler | Group 2 (TDV 1-Dose) Infant/Toddler | Group 3 (TDV 2-Dose) Infant/Toddler | Group 4 (Placebo Control) Infant/Toddler
Number analyzed (Participants) | 29 | 60 | 62 | 32
percentage of participants
  After Vaccination 1, Pain: Any: number analyzed (Participants) | 27 | 54 | 55 | 28
  After Vaccination 1, Pain: Any | 11.1 | 5.6 | 12.7 | 7.1
  After Vaccination 1, Pain: Mild: number analyzed (Participants) | 27 | 54 | 55 | 28
  After Vaccination 1, Pain: Mild | 11.1 | 1.9 | 10.9 | 3.6
  After Vaccination 1, Pain: Moderate: number analyzed (Participants) | 27 | 54 | 55 | 28
  After Vaccination 1, Pain: Moderate | 0 | 3.7 | 1.8 | 3.6
  After Vaccination 1, Erythema: Any: number analyzed (Participants) | 27 | 53 | 55 | 27
  After Vaccination 1, Erythema: Any | 0 | 3.8 | 3.6 | 0
  After Vaccination 1, Erythema (1-2 cm): number analyzed (Participants) | 27 | 53 | 55 | 27
  After Vaccination 1, Erythema (1-2 cm) | 0 | 3.8 | 3.6 | 0
  After Vaccination 1, Swelling: Any: number analyzed (Participants) | 27 | 53 | 55 | 27
  After Vaccination 1, Swelling: Any | 0 | 3.8 | 0 | 0
  After Vaccination 1, Swelling (1-2 cm): number analyzed (Participants) | 27 | 53 | 55 | 27
  After Vaccination 1, Swelling (1-2 cm) | 0 | 3.8 | 0 | 0
  After Vaccination 2, Pain: Any: number analyzed (Participants) | 26 | 53 | 54 | 29
  After Vaccination 2, Pain: Any | 3.8 | 3.8 | 13.0 | 6.9
  After Vaccination 2, Pain: Mild: number analyzed (Participants) | 26 | 53 | 54 | 29
  After Vaccination 2, Pain: Mild | 3.8 | 3.8 | 9.3 | 6.9
  After Vaccination 2, Pain: Moderate: number analyzed (Participants) | 26 | 53 | 54 | 29
  After Vaccination 2, Pain: Moderate | 0 | 0 | 3.7 | 0
  After Vaccination 3, Pain: Any: number analyzed (Participants) | 27 | 56 | 60 | 29
  After Vaccination 3, Pain: Any | 7.4 | 8.9 | 15.0 | 3.4
  After Vaccination 3, Pain: Mild: number analyzed (Participants) | 27 | 56 | 60 | 29
  After Vaccination 3, Pain: Mild | 7.4 | 7.1 | 11.7 | 3.4
  After Vaccination 3, Pain: Moderate: number analyzed (Participants) | 27 | 56 | 60 | 29
  After Vaccination 3, Pain: Moderate | 0 | 1.8 | 1.7 | 0
  After Vaccination 3, Pain: Severe: number analyzed (Participants) | 27 | 56 | 60 | 29
  After Vaccination 3, Pain: Severe | 0 | 0 | 1.7 | 0
  After Vaccination 3, Swelling: Any: number analyzed (Participants) | 27 | 56 | 59 | 29
  After Vaccination 3, Swelling: Any | 0 | 0 | 1.7 | 0
  After Vaccination 3, Swelling (1-2 cm): number analyzed (Participants) | 27 | 56 | 59 | 29
  After Vaccination 3, Swelling (1-2 cm) | 0 | 0 | 1.7 | 0

4. Secondary Outcome: Percentage of Participants With Solicited Local (Injection Site) Adverse Events (AEs) (Diary Recorded) by Severity in the Immunogenicity Subset of Adult/Children Following Each Vaccination
Description: Solicited local injection site reactions were collected by participant diary and graded as [Grade 0 (no pain), 1 (mild: no interference with daily activity), 2 (moderate: interference with daily activity with or without treatment) and 3 (severe: prevents daily activity with or without treatment)]. Erythema and Swelling at injection site were graded as Grade 0 (<25 mm), 1 (mild: ≥25 - ≤ 50 mm), 2 (moderate: > 50 - ≤ 100 mm).
Time Frame: Within 7 days after each vaccination
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Groups:
- Group 1 (TDV 2-Dose) Adult/Children: Participants aged ≥6 years received Takeda's tetravalent dengue vaccine candidate (TDV), 0.5 mL, subcutaneous injection on Days 1 and 91. Placebo-matching, 0.5 mL, subcutaneous injection on Day 365.
- Group 2 (TDV 1-Dose) Adult/Children: Participants aged ≥6 years received Takeda's TDV, 0.5 mL, subcutaneous injection on Day 1. Placebo-matching, 0.5 mL, subcutaneous injection on Days 91 and 365.
- Group 3 (TDV 1-Dose + Booster) Adult/Children: Participants aged ≥6 years received Takeda's TDV, 0.5 mL, subcutaneous injection on Days 1 and 365. Placebo-matching, 0.5 mL, subcutaneous injection on Day 91.
- Group 4 (Placebo Control) Adult/Children: Participant aged ≥6 years received placebo-matching, 0.5 mL, subcutaneous injection on Days 1, 91 and 365.
Arm/Group | Group 1 (TDV 2-Dose) Adult/Children | Group 2 (TDV 1-Dose) Adult/Children | Group 3 (TDV 1-Dose + Booster) Adult/Children | Group 4 (Placebo Control) Adult/Children
Number analyzed (Participants) | 62 | 127 | 129 | 61
percentage of participants
  After Vaccination 1, Pain: Any: number analyzed (Participants) | 60 | 126 | 123 | 57
  After Vaccination 1, Pain: Any | 25.0 | 31.7 | 26.8 | 8.8
  After Vaccination 1, Pain: Mild: number analyzed (Participants) | 60 | 126 | 123 | 57
  After Vaccination 1, Pain: Mild | 23.3 | 28.6 | 22.0 | 7.0
  After Vaccination 1, Pain: Moderate: number analyzed (Participants) | 60 | 126 | 123 | 57
  After Vaccination 1, Pain: Moderate | 1.7 | 2.4 | 4.1 | 1.8
  After Vaccination 1, Pain: Severe: number analyzed (Participants) | 62 | 126 | 123 | 57
  After Vaccination 1, Pain: Severe | 0 | 0.8 | 0.8 | 0
  After Vaccination 1, Erythema: Any: number analyzed (Participants) | 60 | 126 | 122 | 57
  After Vaccination 1, Erythema: Any | 0 | 0.8 | 0 | 0
  After Vaccination 1, Erythema (2.5-5 cm): number analyzed (Participants) | 60 | 126 | 122 | 57
  After Vaccination 1, Erythema (2.5-5 cm) | 0 | 0.8 | 0 | 0
  After Vaccination 1, Swelling: Any: number analyzed (Participants) | 60 | 126 | 122 | 57
  After Vaccination 1, Swelling: Any | 0 | 0 | 0 | 1.8
  After Vaccination 1, Swelling: (2.5-5 cm): number analyzed (Participants) | 60 | 126 | 122 | 57
  After Vaccination 1, Swelling: (2.5-5 cm) | 0 | 0 | 0 | 1.8
  After Vaccination 2, Pain: Any: number analyzed (Participants) | 60 | 116 | 119 | 55
  After Vaccination 2, Pain: Any | 31.7 | 18.1 | 10.9 | 14.5
  After Vaccination 2, Pain: Mild: number analyzed (Participants) | 60 | 116 | 119 | 55
  After Vaccination 2, Pain: Mild | 20.0 | 16.4 | 6.7 | 10.9
  After Vaccination 2, Pain: Moderate: number analyzed (Participants) | 60 | 116 | 119 | 55
  After Vaccination 2, Pain: Moderate | 5.0 | 0 | 4.2 | 1.8
  After Vaccination 2, Pain: Severe: number analyzed (Participants) | 60 | 116 | 119 | 55
  After Vaccination 2, Pain: Severe | 6.7 | 1.7 | 0 | 1.8
  After Vaccination 3, Pain: Any: number analyzed (Participants) | 59 | 115 | 120 | 55
  After Vaccination 3, Pain: Any | 16.9 | 20.0 | 19.2 | 16.4
  After Vaccination 3, Pain: Mild: number analyzed (Participants) | 59 | 115 | 120 | 55
  After Vaccination 3, Pain: Mild | 13.6 | 18.3 | 15.8 | 12.7
  After Vaccination 3, Pain: Moderate: number analyzed (Participants) | 59 | 115 | 120 | 55
  After Vaccination 3, Pain: Moderate | 3.4 | 0 | 3.3 | 3.6
  After Vaccination 3, Pain: Severe: number analyzed (Participants) | 59 | 115 | 120 | 55
  After Vaccination 3, Pain: Severe | 0 | 1.7 | 0 | 0
  After Vaccination 3, Erythema: Any: number analyzed (Participants) | 58 | 115 | 120 | 55
  After Vaccination 3, Erythema: Any | 0 | 0 | 0.8 | 0
  After Vaccination 3, Erythema (2.5-5 cm): number analyzed (Participants) | 58 | 115 | 120 | 55
  After Vaccination 3, Erythema (2.5-5 cm) | 0 | 0 | 0.8 | 0

5. Secondary Outcome: Percentage of Participants With Solicited Systemic Adverse Events (AEs) (Diary Recorded) by Severity in the Immunogenicity Subset of Infant/Toddler Following Each Vaccination
Description: Solicited systemic AEs were collected within 14 days after vaccination using a diary and included drowsiness, graded as 0-behavior as usual, 1-mild: drowsiness easily tolerated, 2-moderate: drowsiness that interferes with normal activity and 3-severe: prevents normal activity with or without treatment; irritability/fussiness, graded as 0-behavior as usual, mild: crying more than usual/no effect on normal activity, moderate: crying more than usual/interferes with normal activity and severe: crying that cannot be comforted/prevents normal; loss of appetite, graded as 0-apetite as usual, mild: eating less than usual/no effect on normal activity, moderate: eating less than usual/interferes with normal activity and severe: not eating at all. A systemic AE of fever (defined as ≥38°C or ≥100.4°F) was derived from a daily temperature reading recorded within 14 days after vaccination. Fever was excluded from the overall count as no severity grading was applied for it.
Time Frame: Within 14 days after each vaccination
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Groups:
- Group 3 (TDV 1-Dose + Booster) Infant/Toddler: Participants aged <6 years received Takeda's TDV, 0.5 mL, subcutaneous injection on Days 1 and 365. Placebo-matching, 0.5 mL, subcutaneous injection on Day 91.
Arm/Group | Group 1 (TDV 2-Dose) Infant/Toddler | Group 2 (TDV 1-Dose) Infant/Toddler | Group 3 (TDV 1-Dose + Booster) Infant/Toddler | Group 4 (Placebo Control) Infant/Toddler
Number analyzed (Participants) | 29 | 60 | 62 | 32
percentage of participants
  After Vaccination 1, Irritability: Any: number analyzed (Participants) | 27 | 54 | 55 | 28
  After Vaccination 1, Irritability: Any | 3.7 | 1.9 | 9.1 | 0
  After Vaccination 1, Irritability: Mild: number analyzed (Participants) | 27 | 54 | 55 | 28
  After Vaccination 1, Irritability: Mild | 3.7 | 0 | 3.6 | 0
  After Vaccination 1, Irritability: Moderate: number analyzed (Participants) | 27 | 54 | 55 | 27
  After Vaccination 1, Irritability: Moderate | 0 | 1.9 | 3.6 | 0
  After Vaccination 1, Irritability: Severe: number analyzed (Participants) | 27 | 54 | 55 | 27
  After Vaccination 1, Irritability: Severe | 0 | 0 | 1.8 | 0
  After Vaccination 1,Drowsiness: Any: number analyzed (Participants) | 27 | 54 | 55 | 28
  After Vaccination 1,Drowsiness: Any | 0 | 7.4 | 7.3 | 7.1
  After Vaccination 1, Drowsiness: Mild: number analyzed (Participants) | 27 | 54 | 55 | 28
  After Vaccination 1, Drowsiness: Mild | 0 | 7.4 | 5.5 | 7.1
  After Vaccination 1, Drowsiness: Moderate: number analyzed (Participants) | 27 | 54 | 55 | 28
  After Vaccination 1, Drowsiness: Moderate | 0 | 0 | 1.8 | 0
  After Vaccination 1,Loss of Appetite:Any: number analyzed (Participants) | 27 | 54 | 55 | 28
  After Vaccination 1,Loss of Appetite:Any | 7.4 | 9.3 | 10.9 | 7.1
  After Vaccination 1,Loss of Appetite: Mild: number analyzed (Participants) | 27 | 54 | 55 | 28
  After Vaccination 1,Loss of Appetite: Mild | 7.4 | 7.4 | 5.5 | 0
  After Vaccination 1, Loss of Appetite: Moderate: number analyzed (Participants) | 27 | 54 | 55 | 28
  After Vaccination 1, Loss of Appetite: Moderate | 0 | 1.9 | 3.6 | 7.1
  After Vaccination 1, Loss of Appetite: Severe: number analyzed (Participants) | 27 | 54 | 55 | 28
  After Vaccination 1, Loss of Appetite: Severe | 0 | 0 | 1.8 | 0
  After Vaccination 1, Fever: Any: number analyzed (Participants) | 25 | 50 | 52 | 27
  After Vaccination 1, Fever: Any | 0 | 6.0 | 5.8 | 3.7
  After Vaccination 1, Fever (38.0 - < 38.5 °C): number analyzed (Participants) | 25 | 50 | 52 | 27
  After Vaccination 1, Fever (38.0 - < 38.5 °C) | 0 | 2.0 | 3.8 | 0
  After Vaccination 1, Fever (38.5 - < 39.0 °C): number analyzed (Participants) | 25 | 50 | 52 | 27
  After Vaccination 1, Fever (38.5 - < 39.0 °C) | 0 | 4.0 | 1.9 | 3.7
  After Vaccination 2, Irritability:Any: number analyzed (Participants) | 26 | 53 | 53 | 28
  After Vaccination 2, Irritability:Any | 15.4 | 1.9 | 1.9 | 10.7
  After Vaccination 2, Irritability: Mild: number analyzed (Participants) | 26 | 53 | 53 | 28
  After Vaccination 2, Irritability: Mild | 15.4 | 1.9 | 1.9 | 10.7
  After Vaccination 2, Drowsiness: Any: number analyzed (Participants) | 26 | 53 | 53 | 28
  After Vaccination 2, Drowsiness: Any | 3.8 | 3.8 | 3.8 | 0
  After Vaccination 2, Drowsiness:Mild: number analyzed (Participants) | 26 | 53 | 53 | 28
  After Vaccination 2, Drowsiness:Mild | 3.8 | 3.8 | 3.8 | 0
  After Vaccination 2, Loss of Appetite: Any: number analyzed (Participants) | 26 | 53 | 53 | 28
  After Vaccination 2, Loss of Appetite: Any | 7.7 | 13.2 | 5.7 | 0
  After Vaccination 2, Loss of Appetite: Mild: number analyzed (Participants) | 26 | 53 | 53 | 28
  After Vaccination 2, Loss of Appetite: Mild | 3.8 | 9.4 | 5.7 | 0
  After Vaccination 2, Loss of Appetite: Moderate: number analyzed (Participants) | 26 | 53 | 53 | 28
  After Vaccination 2, Loss of Appetite: Moderate | 3.8 | 1.9 | 0 | 0
  After Vaccination 2, Loss of Appetite: Severe: number analyzed (Participants) | 26 | 53 | 53 | 28
  After Vaccination 2, Loss of Appetite: Severe | 0 | 1.9 | 0 | 0
  After Vaccination 2, Fever, Any: number analyzed (Participants) | 25 | 52 | 52 | 28
  After Vaccination 2, Fever, Any | 16.0 | 9.6 | 11.5 | 3.6
  After Vaccination 2, Fever (38.0 - < 38.5 °C): number analyzed (Participants) | 25 | 52 | 52 | 28
  After Vaccination 2, Fever (38.0 - < 38.5 °C) | 0 | 3.8 | 5.8 | 0
  After Vaccination 2, Fever (38.5 - < 39.0 °C): number analyzed (Participants) | 25 | 52 | 52 | 28
  After Vaccination 2, Fever (38.5 - < 39.0 °C) | 8.0 | 5.8 | 3.8 | 3.6
  After Vaccination 2, Fever (39.0 - < 39.5 °C): number analyzed (Participants) | 25 | 52 | 52 | 28
  After Vaccination 2, Fever (39.0 - < 39.5 °C) | 4.0 | 0 | 1.9 | 0
  After Vaccination 2, Fever (39.5 - < 40.0 °C): number analyzed (Participants) | 25 | 52 | 52 | 28
  After Vaccination 2, Fever (39.5 - < 40.0 °C) | 4.0 | 0 | 0 | 0
  After Vaccination 3,Irritability: Any: number analyzed (Participants) | 27 | 56 | 59 | 29
  After Vaccination 3,Irritability: Any | 3.7 | 0 | 1.7 | 10.3
  After Vaccination 3, Irritability: Mild: number analyzed (Participants) | 27 | 56 | 59 | 29
  After Vaccination 3, Irritability: Mild | 3.7 | 0 | 0 | 6.9
  After Vaccination 3, Irritability: Moderate: number analyzed (Participants) | 27 | 56 | 59 | 29
  After Vaccination 3, Irritability: Moderate | 0 | 0 | 1.7 | 3.4
  After Vaccination 3,Drowsiness: Any: number analyzed (Participants) | 27 | 56 | 59 | 29
  After Vaccination 3,Drowsiness: Any | 3.7 | 3.6 | 3.4 | 3.4
  After Vaccination 1,Drowsiness: Mild: number analyzed (Participants) | 27 | 56 | 59 | 29
  After Vaccination 1,Drowsiness: Mild | 3.7 | 3.6 | 1.7 | 0
  After Vaccination 1,Drowsiness: Moderate: number analyzed (Participants) | 27 | 56 | 59 | 29
  After Vaccination 1,Drowsiness: Moderate | 0 | 0 | 1.7 | 0
  After Vaccination 3,Drowsiness: Severe: number analyzed (Participants) | 27 | 56 | 59 | 29
  After Vaccination 3,Drowsiness: Severe | 0 | 0 | 0 | 3.4
  After Vaccination 3,Loss of Appetite: Any: number analyzed (Participants) | 27 | 56 | 59 | 29
  After Vaccination 3,Loss of Appetite: Any | 7.4 | 12.5 | 3.4 | 10.3
  After Vaccination 3, Loss of Appetite: Mild: number analyzed (Participants) | 27 | 56 | 59 | 29
  After Vaccination 3, Loss of Appetite: Mild | 3.7 | 7.1 | 3.4 | 6.9
  After Vaccination 3, Loss of Appetite: Moderate: number analyzed (Participants) | 27 | 56 | 59 | 29
  After Vaccination 3, Loss of Appetite: Moderate | 3.7 | 5.4 | 0 | 3.4
  After Vaccination 3, Fever: Any: number analyzed (Participants) | 26 | 55 | 60 | 29
  After Vaccination 3, Fever: Any | 0 | 3.6 | 3.3 | 6.9
  After Vaccination 3, Fever (38.0 - < 38.5 °C): number analyzed (Participants) | 26 | 55 | 60 | 29
  After Vaccination 3, Fever (38.0 - < 38.5 °C) | 0 | 0 | 1.7 | 3.4
  After Vaccination 3, Fever (38.5 - < 39.0 °C): number analyzed (Participants) | 26 | 55 | 60 | 29
  After Vaccination 3, Fever (38.5 - < 39.0 °C) | 0 | 1.8 | 1.7 | 0
  After Vaccination 3, Fever (39.0 - < 39.5 °C): number analyzed (Participants) | 26 | 55 | 60 | 29
  After Vaccination 3, Fever (39.0 - < 39.5 °C) | 0 | 1.8 | 0 | 3.4

6. Secondary Outcome: Percentage of Participants With Solicited Systemic Adverse Events (AEs) (Diary Recorded) by Severity in the Immunogenicity Subset of Adult/Children Following Each Vaccination
Description: Solicited systemic AEs were collected by participants within 14 days after vaccination and included headache, asthenia, malaise, myalgia and fever. Severity scales for headache were none, mild: no interference with daily activity, moderate: interference with daily activity with or without treatment and severe: prevents normal activity with or without treatment. Severity scales for others were none, mild: no interference with daily activity, moderate: interference with daily activity and severe: prevents daily activity. A systemic AE of fever (defined as ≥38°C or ≥100.4°F) was derived from a daily temperature reading recorded within 14 days after vaccination. Fever was excluded from the overall count as no severity grading was applied for it.
Time Frame: Within 14 days after each vaccination
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Groups:
- Group 4 (Placebo Control) Adult/Children: Participants aged ≥6 years received placebo-matching, 0.5 mL, subcutaneous injection on Days 1, 91 and 365.
Arm/Group | Group 1 (TDV 2-Dose) Adult/Children | Group 2 (TDV 1-Dose) Adult/Children | Group 3 (TDV 1-Dose + Booster) Adult/Children | Group 4 (Placebo Control) Adult/Children
Number analyzed (Participants) | 62 | 127 | 129 | 61
percentage of participants
  After Vaccination 1, Headache: Any: number analyzed (Participants) | 60 | 126 | 123 | 57
  After Vaccination 1, Headache: Any | 20.0 | 23.8 | 16.3 | 21.1
  After Vaccination 1, Headache: Mild: number analyzed (Participants) | 60 | 126 | 123 | 57
  After Vaccination 1, Headache: Mild | 16.7 | 20.6 | 13.0 | 14.0
  After Vaccination 1, Headache: Moderate: number analyzed (Participants) | 60 | 126 | 123 | 57
  After Vaccination 1, Headache: Moderate | 3.3 | 2.4 | 1.6 | 5.3
  After Vaccination 1, Headache: Severe: number analyzed (Participants) | 60 | 126 | 123 | 57
  After Vaccination 1, Headache: Severe | 0 | 0.8 | 1.6 | 1.8
  After Vaccination 1, Asthenia: Any: number analyzed (Participants) | 60 | 126 | 123 | 57
  After Vaccination 1, Asthenia: Any | 5.0 | 11.1 | 7.3 | 7.0
  After Vaccination 1, Asthenia: Mild: number analyzed (Participants) | 60 | 126 | 123 | 57
  After Vaccination 1, Asthenia: Mild | 3.3 | 10.3 | 4.9 | 3.5
  After Vaccination 1, Asthenia: Moderate: number analyzed (Participants) | 60 | 126 | 123 | 57
  After Vaccination 1, Asthenia: Moderate | 1.7 | 0.8 | 1.6 | 3.5
  After Vaccination 1, Asthenia: Severe: number analyzed (Participants) | 60 | 126 | 123 | 57
  After Vaccination 1, Asthenia: Severe | 0 | 0 | 0.8 | 0
  After Vaccination 1, Malaise: Any: number analyzed (Participants) | 60 | 126 | 123 | 57
  After Vaccination 1, Malaise: Any | 8.3 | 14.3 | 8.9 | 10.5
  After Vaccination 1, Malaise: Mild: number analyzed (Participants) | 60 | 126 | 123 | 57
  After Vaccination 1, Malaise: Mild | 6.7 | 13.5 | 7.3 | 8.8
  After Vaccination 1, Malaise: Moderate: number analyzed (Participants) | 60 | 126 | 123 | 57
  After Vaccination 1, Malaise: Moderate | 1.7 | 0.8 | 0.8 | 0
  After Vaccination 1, Malaise: Severe: number analyzed (Participants) | 60 | 126 | 123 | 57
  After Vaccination 1, Malaise: Severe | 0 | 0 | 0.8 | 1.8
  After Vaccination 1, Myalgia: Any: number analyzed (Participants) | 60 | 126 | 123 | 57
  After Vaccination 1, Myalgia: Any | 10.0 | 20.6 | 11.4 | 7.0
  After Vaccination 1, Myalgia: Mild: number analyzed (Participants) | 60 | 126 | 123 | 57
  After Vaccination 1, Myalgia: Mild | 8.3 | 18.3 | 10.6 | 7.0
  After Vaccination 1, Myalgia: Moderate: number analyzed (Participants) | 60 | 126 | 123 | 57
  After Vaccination 1, Myalgia: Moderate | 1.7 | 2.4 | 0 | 0
  After Vaccination 1, Myalgia: Severe: number analyzed (Participants) | 60 | 126 | 123 | 57
  After Vaccination 1, Myalgia: Severe | 0 | 0 | 0.8 | 0
  After Vaccination 1, Fever: Any: number analyzed (Participants) | 51 | 119 | 110 | 51
  After Vaccination 1, Fever: Any | 5.9 | 2.5 | 4.5 | 5.9
  After Vaccination 1, Fever: 38.0 - < 38.5 °C: number analyzed (Participants) | 51 | 119 | 110 | 51
  After Vaccination 1, Fever: 38.0 - < 38.5 °C | 2.0 | 1.7 | 0 | 2.0
  After Vaccination 1, Fever: 38.5 - < 39.0 °C: number analyzed (Participants) | 51 | 119 | 110 | 51
  After Vaccination 1, Fever: 38.5 - < 39.0 °C | 2.0 | 0 | 1.8 | 3.9
  After Vaccination 1, Fever: 39.0 - < 39.5 °C: number analyzed (Participants) | 51 | 119 | 110 | 51
  After Vaccination 1, Fever: 39.0 - < 39.5 °C | 2.0 | 0.8 | 0.9 | 0
  After Vaccination 1, Fever: 39.5 - < 40.0 °C: number analyzed (Participants) | 51 | 119 | 110 | 51
  After Vaccination 1, Fever: 39.5 - < 40.0 °C | 0 | 0 | 1.8 | 0
  After Vaccination 2, Headache: Any: number analyzed (Participants) | 59 | 115 | 118 | 55
  After Vaccination 2, Headache: Any | 18.6 | 9.6 | 6.8 | 16.4
  After Vaccination 2, Headache: Mild: number analyzed (Participants) | 59 | 115 | 118 | 55
  After Vaccination 2, Headache: Mild | 11.9 | 7.8 | 4.2 | 12.7
  After Vaccination 2, Headache: Moderate: number analyzed (Participants) | 59 | 115 | 118 | 55
  After Vaccination 2, Headache: Moderate | 5.1 | 0.9 | 2.5 | 1.8
  After Vaccination 2, Headache: Severe: number analyzed (Participants) | 59 | 115 | 118 | 55
  After Vaccination 2, Headache: Severe | 1.7 | 0.9 | 0 | 1.8
  After Vaccination 2, Asthenia: Any: number analyzed (Participants) | 59 | 115 | 118 | 55
  After Vaccination 2, Asthenia: Any | 8.5 | 7.8 | 4.2 | 3.6
  After Vaccination 2, Asthenia: Mild: number analyzed (Participants) | 59 | 115 | 118 | 55
  After Vaccination 2, Asthenia: Mild | 5.1 | 7.0 | 2.5 | 3.6
  After Vaccination 2, Asthenia: Moderate: number analyzed (Participants) | 59 | 115 | 118 | 55
  After Vaccination 2, Asthenia: Moderate | 1.7 | 0 | 1.7 | 0
  After Vaccination 2, Asthenia: Severe: number analyzed (Participants) | 59 | 115 | 118 | 55
  After Vaccination 2, Asthenia: Severe | 1.7 | 0.9 | 0 | 0
  After Vaccination 2, Malaise: Any: number analyzed (Participants) | 59 | 115 | 118 | 55
  After Vaccination 2, Malaise: Any | 15.3 | 8.7 | 6.8 | 9.1
  After Vaccination 2, Malaise: Mild: number analyzed (Participants) | 59 | 115 | 118 | 55
  After Vaccination 2, Malaise: Mild | 10.2 | 6.1 | 4.2 | 7.3
  After Vaccination 2, Malaise: Moderate: number analyzed (Participants) | 59 | 115 | 118 | 55
  After Vaccination 2, Malaise: Moderate | 3.4 | 1.7 | 1.7 | 0
  After Vaccination 2, Malaise: Severe: number analyzed (Participants) | 59 | 115 | 118 | 55
  After Vaccination 2, Malaise: Severe | 1.7 | 0.9 | 0.8 | 1.8
  After Vaccination 2, Myalgia: Any: number analyzed (Participants) | 59 | 115 | 118 | 55
  After Vaccination 2, Myalgia: Any | 16.9 | 5.2 | 5.9 | 5.5
  After Vaccination 2, Myalgia: Mild: number analyzed (Participants) | 59 | 115 | 118 | 55
  After Vaccination 2, Myalgia: Mild | 10.2 | 5.2 | 2.5 | 5.5
  After Vaccination 2, Myalgia: Moderate: number analyzed (Participants) | 59 | 115 | 118 | 55
  After Vaccination 2, Myalgia: Moderate | 3.4 | 0 | 2.5 | 0
  After Vaccination 2, Myalgia: Severe: number analyzed (Participants) | 59 | 115 | 118 | 55
  After Vaccination 2, Myalgia: Severe | 3.4 | 0 | 0.8 | 0
  After Vaccination 2, Fever: Any: number analyzed (Participants) | 51 | 104 | 110 | 49
  After Vaccination 2, Fever: Any | 2.0 | 2.9 | 2.7 | 4.1
  After Vaccination 2, Fever: 38.0 - < 38.5 °C: number analyzed (Participants) | 51 | 104 | 110 | 49
  After Vaccination 2, Fever: 38.0 - < 38.5 °C | 2.0 | 1.0 | 0.9 | 0
  After Vaccination 2, Fever: 38.5 - < 39.0 °C: number analyzed (Participants) | 51 | 104 | 110 | 49
  After Vaccination 2, Fever: 38.5 - < 39.0 °C | 0 | 1.0 | 0.9 | 2.0
  After Vaccination 2, Fever: 39.5 - < 40.0 °C: number analyzed (Participants) | 51 | 104 | 110 | 49
  After Vaccination 2, Fever: 39.5 - < 40.0 °C | 0 | 1.0 | 0.9 | 2.0
  After Vaccination 3, Headache: Any: number analyzed (Participants) | 59 | 115 | 120 | 55
  After Vaccination 3, Headache: Any | 10.2 | 11.3 | 7.5 | 7.3
  After Vaccination 3, Headache: Mild: number analyzed (Participants) | 59 | 115 | 120 | 55
  After Vaccination 3, Headache: Mild | 10.2 | 7.8 | 5.8 | 5.5
  After Vaccination 3, Headache: Moderate: number analyzed (Participants) | 59 | 115 | 120 | 55
  After Vaccination 3, Headache: Moderate | 0 | 1.7 | 1.7 | 0
  After Vaccination 3, Headache: Severe: number analyzed (Participants) | 59 | 115 | 120 | 55
  After Vaccination 3, Headache: Severe | 0 | 1.7 | 0 | 1.8
  After Vaccination 3, Asthenia: Any: number analyzed (Participants) | 59 | 115 | 120 | 55
  After Vaccination 3, Asthenia: Any | 6.8 | 7.0 | 2.5 | 7.3
  After Vaccination 3, Asthenia: Mild: number analyzed (Participants) | 59 | 115 | 120 | 55
  After Vaccination 3, Asthenia: Mild | 6.8 | 5.2 | 2.5 | 7.3
  After Vaccination 3, Asthenia: Moderate: number analyzed (Participants) | 59 | 115 | 120 | 55
  After Vaccination 3, Asthenia: Moderate | 0 | 0.9 | 0 | 0
  After Vaccination 3, Asthenia: Severe: number analyzed (Participants) | 59 | 115 | 120 | 55
  After Vaccination 3, Asthenia: Severe | 0 | 0.9 | 0 | 0
  After Vaccination 3, Malaise: Any: number analyzed (Participants) | 59 | 115 | 120 | 55
  After Vaccination 3, Malaise: Any | 5.1 | 7.8 | 8.3 | 3.6
  After Vaccination 3, Malaise: Mild: number analyzed (Participants) | 59 | 115 | 120 | 55
  After Vaccination 3, Malaise: Mild | 3.4 | 5.2 | 5.8 | 1.8
  After Vaccination 3, Malaise: Moderate: number analyzed (Participants) | 59 | 115 | 120 | 55
  After Vaccination 3, Malaise: Moderate | 0 | 0.9 | 1.7 | 1.8
  After Vaccination 3, Malaise: Severe: number analyzed (Participants) | 59 | 115 | 120 | 55
  After Vaccination 3, Malaise: Severe | 1.7 | 1.7 | 0.8 | 0
  After Vaccination 3, Myalgia: Any: number analyzed (Participants) | 59 | 115 | 120 | 55
  After Vaccination 3, Myalgia: Any | 6.8 | 11.3 | 8.3 | 5.5
  After Vaccination 3, Myalgia: Mild: number analyzed (Participants) | 59 | 115 | 120 | 55
  After Vaccination 3, Myalgia: Mild | 5.1 | 9.6 | 5.8 | 5.5
  After Vaccination 3, Myalgia: Moderate: number analyzed (Participants) | 59 | 115 | 120 | 55
  After Vaccination 3, Myalgia: Moderate | 0 | 0.9 | 1.7 | 0
  After Vaccination 3, Myalgia: Severe: number analyzed (Participants) | 59 | 115 | 120 | 55
  After Vaccination 3, Myalgia: Severe | 1.7 | 0.9 | 0.8 | 0
  After Vaccination 3, Fever: Any: number analyzed (Participants) | 56 | 106 | 115 | 51
  After Vaccination 3, Fever: Any | 1.8 | 1.9 | 1.7 | 2.0
  After Vaccination 3, Fever: 38.0 - < 38.5 °C: number analyzed (Participants) | 56 | 106 | 115 | 51
  After Vaccination 3, Fever: 38.0 - < 38.5 °C | 0 | 1.9 | 0.9 | 2.0
  After Vaccination 3, Fever: 38.5 - < 39.0 °C: number analyzed (Participants) | 56 | 106 | 115 | 51
  After Vaccination 3, Fever: 38.5 - < 39.0 °C | 0 | 0 | 0.9 | 0
  After Vaccination 3, Fever: 39.0 - < 39.5 °C: number analyzed (Participants) | 56 | 106 | 115 | 51
  After Vaccination 3, Fever: 39.0 - < 39.5 °C | 1.8 | 0 | 0 | 0

7. Secondary Outcome: Percentage of Participants With Any Unsolicited Adverse Events (AEs) in the Immunogenicity Subset Following Each Vaccination
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment.
Time Frame: Within 28 days after each vaccination
Population: Safety Analysis Set included all participants who received at least 1 dose of trial vaccine. Safety Set included only participants from Immunogenicity Subset with data available for analyses. Number analyzed is number of participants with data available after each vaccination.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1 (TDV 2-Dose) | Group 2 (TDV 1-Dose) | Group 3 (TDV 1-Dose + Booster) | Group 4 (Placebo Control)
Number analyzed (Participants) | 91 | 187 | 191 | 93
percentage of participants
  After Vaccination 1 | 19.8 | 20.3 | 19.4 | 21.5
  After Vaccination 2: number analyzed (Participants) | 90 | 176 | 181 | 87
  After Vaccination 2 | 12.2 | 10.2 | 11.0 | 16.1
  After Vaccination 3: number analyzed (Participants) | 88 | 172 | 179 | 84
  After Vaccination 3 | 6.8 | 12.8 | 10.1 | 9.5

8. Secondary Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Description: An SAE was defined as any untoward medical occurrence or effect that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically important due to other reasons than the above-mentioned criteria.
Time Frame: From first vaccination through end of study (Day 1460)
Population: Safety Analysis Set included all participants who received at least 1 dose of trial vaccine.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1 (TDV 2-Dose) | Group 2 (TDV 1-Dose) | Group 3 (TDV 1-Dose + Booster) | Group 4 (Placebo Control)
Number analyzed (Participants) | 200 | 398 | 998 | 198
percentage of participants | 5.0 | 4.5 | 6.5 | 5.1

9. Secondary Outcome: Percentage of Participants With Febrile Episodes of Virologically Confirmed Dengue With Onset 30 Days Post-first Vaccination
Description: Participants with febrile illness (defined as temperature ≥ 38°C on 2 consecutive days) were evaluated for dengue. A dengue infection was considered virologically confirmed by either positive polymerase chain reaction (PCR) or NS1 enzyme-linked immunosorbent assay (ELISA). Virologically confirmed dengue with onset 30 days after first vaccination within each group.
Time Frame: From 30 days post-first vaccination through end of study (Day 1460)
Population: Safety Analysis Set included all participants who received at least 1 dose of trial vaccine.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1 (TDV 2-Dose) | Group 2 (TDV 1-Dose) | Group 3 (TDV 1-Dose + Booster) | Group 4 (Placebo Control)
Number analyzed (Participants) | 200 | 398 | 998 | 198
percentage of participants | 3.5 | 2.0 | 2.2 | 6.6

ADVERSE EVENTS:
Time Frame: All-Cause Mortality and Serious adverse events: From first vaccination (Day 1) through end of study (Day 540); Other adverse events: From any vaccination (Day 1, Day 91, and Day 365) up to 28 days post vaccination.
Description: Safety Analysis Set included all participants who received at least 1 dose of trial vaccine. Data for other (non-serious) adverse events is reported for participants from Immunogenicity Subset with available data for analyses.
Arm/Group | Group 1 (TDV 2-Dose) | Group 2 (TDV 1-Dose) | Group 3 (TDV 1-Dose + Booster) | Group 4 (Placebo Control)
All-Cause Mortality (participants affected / at risk) | 0/200 | 1/398 | 1/998 | 0/198
Serious Adverse Events (participants affected / at risk) | 10/200 | 18/398 | 65/998 | 10/198
Other Adverse Events (participants affected / at risk) | 17/91 | 43/187 | 41/191 | 22/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (TDV 2-Dose) (N=200) | Group 2 (TDV 1-Dose) (N=398) | Group 3 (TDV 1-Dose + Booster) (N=998) | Group 4 (Placebo Control) (N=198)
Immune Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Ocular Myasthenia (Eye disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus Paralytic (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Volvulus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dehiscence (General disorders) | 0 | 0 | 1 | 0
Food Allergy (Immune system disorders) | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Amoebic Dysentery (Infections and infestations) | 1 | 1 | 5 | 1
Gastroenteritis (Infections and infestations) | 0 | 2 | 5 | 1
Appendicitis (Infections and infestations) | 2 | 0 | 4 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 5 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 4 | 0
Abscess Limb (Infections and infestations) | 0 | 0 | 1 | 1
Ascariasis (Infections and infestations) | 0 | 1 | 1 | 0
Dengue Fever (Infections and infestations) | 0 | 1 | 1 | 0
Scarlet Fever (Infections and infestations) | 0 | 0 | 2 | 0
Amoebiasis (Infections and infestations) | 0 | 0 | 1 | 0
Appendicitis Perforated (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Burkholderia Cepacia Complex Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Encephalomyelitis (Infections and infestations) | 0 | 1 | 0 | 0
Endometritis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis Rotavirus (Infections and infestations) | 0 | 0 | 1 | 0
Hepatitis A (Infections and infestations) | 0 | 0 | 1 | 0
Infectious Colitis (Infections and infestations) | 0 | 0 | 1 | 0
Nasal Abscess (Infections and infestations) | 0 | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 0 | 1 | 0
Peritonsillar Abscess (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 1 | 0 | 0
Pulmonary Tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Septic Shock (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0
Tooth Abscess (Infections and infestations) | 0 | 0 | 1 | 0
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 0
Head Injury (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0
Multiple Injuries (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0
Abdominal Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Arthropod Sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Burns Second Degree (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Aneurysmal Bone Cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Teratoma Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 2 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0
Generalised Tonic-Clonic (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Relapsing-Remitting Multiple Sclerosis (Nervous system disorders) | 0 | 1 | 0 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Premature Baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Glomerulonephritis Acute (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nephritic Syndrome (Renal and urinary disorders) | 0 | 0 | 0 | 1
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Ovarian Cyst Torsion (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Asthmatic Crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Homicide (Social circumstances) | 0 | 0 | 1 | 0
Finger Amputation (Surgical and medical procedures) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (TDV 2-Dose) (N=91) | Group 2 (TDV 1-Dose) (N=187) | Group 3 (TDV 1-Dose + Booster) (N=191) | Group 4 (Placebo Control) (N=93)
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 2 | 2
Vomiting (Gastrointestinal disorders) | 1 | 3 | 0 | 3
Pyrexia (General disorders) | 2 | 1 | 2 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 2 | 2
Nasopharyngitis (Infections and infestations) | 10 | 25 | 21 | 10
Viral Infection (Infections and infestations) | 1 | 4 | 4 | 2
Bronchitis (Infections and infestations) | 0 | 4 | 3 | 0
Tonsillitis (Infections and infestations) | 2 | 3 | 2 | 0
Parasitic Gastroenteritis (Infections and infestations) | 2 | 0 | 1 | 2
Headache (Nervous system disorders) | 1 | 2 | 5 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 7 | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-05-31): https://cdn.clinicaltrials.gov/large-docs/66/NCT02302066/SAP_000.pdf
  • Study Protocol (2016-07-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT02302066/Prot_001.pdf